CLINICAL TRIAL: NCT06379425
Title: Impact of Preoperative Opioid-free Multimodal Analgesia on Time to Trial of Void in Ambulatory Urogynecologic Surgeries: A Randomized Controlled Trial
Brief Title: Impact of Preoperative Opioid-free Multimodal Analgesia on Time to Trial of Void in Ambulatory Urogynecologic Surgeries
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 23-0050
Record Dates: First submitted 2024-04-03; First posted 2024-04-23 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Pain, Postoperative; Postoperative Pain, Acute
MeSH Terms: conditions — Pain, Postoperative | interventions — Acetaminophen; Celecoxib; Gabapentin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard of Care (SOC) (acetaminophen) (Active Comparator): one time dose of 1000mg acetaminophen orally
  Interventions: Drug: Acetaminophen
- Standard of Care (SOC) (acetaminophen) and investigational product (celecoxib + gabapentin) (Experimental): one time dose of 1000mg acetaminophen orally combined with 400mg celecoxib orally, and 300mg gabapentin orally
  Interventions: Drug: Acetaminophen; Drug: Celecoxib; Drug: Gabapentin

INTERVENTIONS:
Drug: Acetaminophen — Will add additional medications celecoxib and gabapentin to acetaminophen preoperatively prior to patient surgery
Drug: Celecoxib — Will add additional medications celecoxib and gabapentin to acetaminophen preoperatively prior to patient surgery
  Arms: Standard of Care (SOC) (acetaminophen) and investigational product (celecoxib + gabapentin)
Drug: Gabapentin — Will add additional medications celecoxib and gabapentin to acetaminophen preoperatively prior to patient surgery
  Arms: Standard of Care (SOC) (acetaminophen) and investigational product (celecoxib + gabapentin)

SUMMARY:
This is a double-arm randomized control trial evaluating the impact of preoperative opioid-free analgesia on time to trial of void in ambulatory urogynecologic surgeries. The investigators hypothesize that receipt of acetaminophen, celecoxib and gabapentin preoperatively versus acetaminophen alone will reduce the time to trial of void in patients undergoing same-day minor urogynecologic procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. All female patients over 18 years of age from the Northwell Health urogynecology offices in Bay Shore, Syosset, and Huntington, NY who are undergoing transvaginal minor urogynecologic surgery (midurethral sling, periurethral bulking injections, anterior repair, posterior repair, and perineorrhaphy) at South Shore Surgery Center
4. In good general health as evidenced by medical history
5. Ability to take oral medication and be willing to adhere to the study intervention
6. Patients may be English or Spanish-speaking and must be able to provide informed consent

Exclusion Criteria:

1. Pregnancy or lactation
2. Younger than age 18
3. Known allergic reactions to acetaminophen, celecoxib or gabapentin or any components within the medication formulation
4. Patients with Myasthenia Gravis, renal disease with CrCl < 50, seizure disorder, substance use disorder, anaphylaxis and angioedema to gabapentin, Drug reaction with Eosinophilia and Systemic Symptoms (DRESS), driving impairment, increased seizures suicidal behavior and respiratory depression.
5. Patients with a , history of asthma, urticaria, or other allergic type reactions after taking aspirin or other NSAIDS or DRESS, history of gastric bypass surgery, heart failure, active GI ulcer, active GI bleeding, inflammatory bowel disease, cerebrovascular bleeding, liver impairment/hepatic disease, hyperkalemia.
6. Patients with compromised renal function who are notable to receive NSAIDs
7. Patients with significant cardiovascular disease, such as patients with heart failure
8. Patient with recent evidence of worsening fluid retention
9. Both non-English and non-Spanish speaking patients
10. Urogynecologic surgeries for apical repair (sacrocolpopexy, uterosacral ligament suspension, sacrospinous ligament suspension, colpocleisis)
11. Current use of illicit substances (cocaine, non-prescription opioids, marijuana)
12. Current use of gabapentin as home medication

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Time to initiation of active trial of void | through study completion, an average of 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Northwell Health South Shore Surgery Center, Bay Shore, New York, United States